CLINICAL TRIAL: NCT00270660
Title: A Cross Sectional Study of Clinicopathologic Behaviour of Primary, Secondary and Mixed Types of Atticoantral Chronic Otitis Media
Brief Title: A Study of the Clinicopathologic Behaviour of the Different Types of Unsafe Chronic Otitis Media
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karnataka Institute of Medical Sciences (Other)
Other Study IDs: M06a/2003-04
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2005-12

CONDITIONS: Chronic Otitis Media; Cholesteatoma
Keywords: retraction pockets ear; unsafe otitis media; otitis media complications
MeSH Terms: conditions — Cholesteatoma | interventions — Biopsy; Hearing

STUDY DESIGN:
Time Perspective: Other

INTERVENTIONS:
Behavioral: biopsy, audiometry, ET function test, ear swab culture, DNE

SUMMARY:
The purpose of the study is to study the clinicopathologic behaviour of the 3 dangerous types of chronic otitis media that are prone for complications. In which type are the complications more common? Which type gives rise to more hearing loss? How does the disease process in the 3 types evolve? should the 3 types of otitis media be managed differently?

DETAILED DESCRIPTION:
Design: prospective cross sectional study setting: tertiary referral medical college hospital No of groups: 3 group 1: primary acquired atticoantral disease group 2: secondary acquired atticoantral disease group 3: mixed atticoantral disease

Interventions:

1. Diagnostic nasal endoscopy
2. Eustachian tube function tests
3. Pure tone audiometry
4. biopsy of middle ear mucosa
5. culture and sensitivity of ear discharge

ELIGIBILITY:
Inclusion Criteria:1. Atticoantral chronic otitis media 2. complicated unsafe otitis media 3. Otitis media with cholesteatoma, polyp, granulation tissue 4. Ear with retraction pockets leading to attic -

Exclusion Criteria:

1. tubotympanic otitis media alone
2. otitis media with effusion
3. Acute otitis media -

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192
Dates: Start 2003-07; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Vikram K Bhat, MS, DNB., Principal Investigator — Karnataka Institute of Medical Sciences, Hubli, India; Khaja Naseeruddin, MS, DLO., Study Director — Vijayanagar Institute of Medical Sciences, Bellary, India
Locations (1):
- Department of ENT, KIMS, Hubli, Karnataka, India